CLINICAL TRIAL: NCT03054389
Title: Non-Interventional Study to Capture the Patient Experience on Gene Therapy for Hemophilia Within the AskBio009-101 Study Through Patient and Investigator Interviews
Status: Completed | Type: Observational
Sponsor: Baxalta now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Other Study IDs: 001601
Record Dates: First submitted 2017-02-13; First posted 2017-02-15 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Hemophilia B
MeSH Terms: conditions — Hemophilia B

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Participants/ Patients: Participants/ Patients from the AskBio009-101 Study
  Interventions: Other: Qualitative Interview - Participants/ Patients
- Investigators and Study Coordinators: Investigators and Study Coordinators from the AskBio009-101 Study
  Interventions: Other: Qualitative Interview - Investigators and Study Coordinators

INTERVENTIONS:
Other: Qualitative Interview - Participants/ Patients — Qualitative interviews to understand the patient experience with the AskBio009-101 Study - Participants/ Patients
  Groups: Participants/ Patients
Other: Qualitative Interview - Investigators and Study Coordinators — Qualitative interviews to understand the patient experience with the AskBio009-101 Study - Investigators and Study Coordinators
  Groups: Investigators and Study Coordinators

SUMMARY:
The purpose of this study is to seek to understand the patient's perspective around deciding to participate in a clinical trial for a Hemophilia therapy

ELIGIBILITY:
Inclusion criteria for patients:

* Were screened and consented for the AskBio009-101study at any point in time
* Are able to speak and understand English
* Are between ages of 18 and 75
* Are physically able to participate in a one-hour phone interview
* Consented into this study independently of the AskBio009-101 study

Exclusion criteria for patients:

- N/A

Inclusion criteria for investigators and coordinators:

* Worked at a site as an investigator or study coordinator that consented a patient into the
* AskBio009-101 trial at any point in time, including those that no longer work at a AskBio009-101 site
* Are able to speak and understand English
* Are between ages of 18 and 75
* Are physically able to participate in a one-hour phone interview

Exclusion criteria for investigators and coordinators:

- Not directly involved in the consent process at the gene therapy site

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Investigators, Study Coordinators, and Participants from the AskBio009-101 Study
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2017-03-31 (Actual); Primary Completion 2017-06-06 (Actual); Study Completion 2017-06-06 (Actual)

PRIMARY OUTCOMES:
Interview - AskBio009-101 Study - Participants/ Patients | Approximately 1 hour
  Qualitative telephone interviews to understand the patient experience with the AskBio009-101 Study - Participant/ Patient Interview
Interview - AskBio009-101 Study - Investigators and Study Coordinators | Approximately 1 hour
  Qualitative telephone interviews to understand the patient experience with the AskBio009-101 Study - Investigators and Study Coordinators Interview

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- QuintilesIMS, Cambridge, Massachusetts, United States